CLINICAL TRIAL: NCT06320249
Title: Rotation-traction Manipulation of Different Treatment Frequency in Cervical Radiculopathy: A Multicenter Randomized Controlled Trial
Brief Title: Rotation-traction Manipulation of Different Treatment Frequency in Cervical Radiculopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other)
Collaborators: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Affiliated Hospital of Changchun University of Chinese Medicine (Other); Dongzhimen Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WJYY-XZKT-2023-05
Record Dates: First submitted 2024-02-24; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cervical Radiculopathy
Keywords: Rotation-traction manipulation; Cervical radiculopathy; Treatment frequency; Dose effect; Randomized controlled trial
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study did not implement blinding for the manipulative therapists and participants. However, blinding procedures were employed for the outcome assessors and data analysts, meaning that they remained unaware of the group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The high-frequency manipulation group (Experimental): In the high-frequency manipulation group, patients will undergo rotation-traction manipulation three times weekly. A total of 12 treatments for four weeks.
  Interventions: Other: High-frequency rotation-traction manipulation
- The low-frequency manipulation group (Experimental): In the low-frequency manipulation group, patients will undergo rotation-traction manipulation once time weekly. A total of 4 treatments for four weeks.
  Interventions: Other: Low-frequency rotation-traction manipulation
- The cervical traction group (Active Comparator): The cervical traction group will be subjected to cervical traction three times a week. A total of 12 treatments for four weeks.
  Interventions: Other: Cervical traction

INTERVENTIONS:
Other: High-frequency rotation-traction manipulation — The procedure for rotation-traction manipulation is as follows: The patient is seated, and their neck is allowed to relax. The physician applies massage techniques to relax the muscles around the neck area for approximately 5 to 10 minutes. The patient is then instructed to rotate their head horizontally, flex it, and then rotate it again to its maximum limit while maintaining a sense of fixation. The physician supports the patient's chin with their elbow and gently pulls upward for 3 to 5 seconds. The patient is then asked to fully relax, and the physician applies a quick, short upward traction with the elbow, which may result in audible sounds. Subsequently, massage techniques are applied to further relax the muscles around the neck and shoulders, with each session lasting approximately 10 to 15 minutes. In the high-frequency manipulation group, patients will undergo rotation-traction manipulation three times weekly. A total of 12 treatments for four weeks.
  Arms: The high-frequency manipulation group
Other: Low-frequency rotation-traction manipulation — The procedure for rotation-traction manipulation is as follows: The patient is seated, and their neck is allowed to relax. The physician applies massage techniques to relax the muscles around the neck area for approximately 5 to 10 minutes. The patient is then instructed to rotate their head horizontally, flex it, and then rotate it again to its maximum limit while maintaining a sense of fixation. The physician supports the patient's chin with their elbow and gently pulls upward for 3 to 5 seconds. The patient is then asked to fully relax, and the physician applies a quick, short upward traction with the elbow, which may result in audible sounds. Subsequently, massage techniques are applied to further relax the muscles around the neck and shoulders, with each session lasting approximately 10 to 15 minutes. In the low-frequency manipulation group, patients will undergo rotation-traction manipulation once time weekly. A total of 4 treatments for four weeks.
  Arms: The low-frequency manipulation group
Other: Cervical traction — The procedure for cervical traction is as follows: The patient assumes a sitting position, and a cervical traction device with a chin strap is applied. The patient is instructed to slightly flex their head forward, approximately 10-15 degrees, based on their comfort level and symptom relief. Traction force starts at 3 kg and increases gradually in increments of 0.5 kg, with a maximum weight not exceeding 6 kg. The cervical traction group will be subjected to cervical traction three times a week. A total of 12 treatments for four weeks.
  Arms: The cervical traction group

SUMMARY:
The evidence for different frequencies of rotation-traction manipulation treatment in cervical radiculopathy is insufficient. This study determined whether 3 sessions per week of rotation-traction manipulation treatment are superior to 1 session per week for symptomatic outcomes in cervical radiculopathy based on a multicenter randomized controlled trial.

DETAILED DESCRIPTION:
This study, slated to be conducted across four sub-centers, including the Wangjing Hospital of the China Academy of Chinese Medical Sciences, aims to recruit 216 patients diagnosed with cervical radiculopathy. Employing a central randomization method, participants will be stratified into three groups: high-frequency manipulation, low-frequency manipulation, and cervical traction.

In the high-frequency manipulation group, patients will undergo rotation-traction manipulation three times weekly, while the low-frequency manipulation group will receive the same intervention once a week. The cervical traction group will be subjected to cervical traction three times a week. Each group will undergo 4-week treatment with a subsequent 16-week follow-up, resulting in a total study duration of 20 weeks.

Outcomes' assessments will be conducted at seven specific time points: baseline, 2 weeks after treatment, 4 weeks after treatment, and during follow-up at weeks 4, 8, 12, and 16. Outcomes include scores from the Visual Analog Scale (VAS) for pain, VAS for numbness, Neck Disability Index (NDI), Short Form-12 (SF-12) health survey, and monitoring of adverse reactions. Following the first treatment session and 4 weeks after treatment, Expectation Treatment Credibility Scale (ETCS) will be appraised. Furthermore, the study will record the overall cost incurred by each group after 4 weeks of treatment and the recurrence rates during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Conforming to the diagnostic criteria outlined in the 2010 North American Spine Society "An evidence-based clinical guideline for the diagnosis and treatment of cervical radiculopathy from degenerative disorders".
2. Aged between 40 and 65 years.
3. VAS score ≥ 4 points.
4. Duration of the condition ≤ 5 years.
5. Voluntary signature of informed consent form.

Exclusion Criteria:

1. Combined with other types of cervical spondylosis.
2. Suspected or confirmed cases of cervical spine or intraspinal tumor, or intracranial tumor.
3. Patients with unclear diagnosis of spinal injury or symptoms of spinal cord injury.
4. Patients with developmental spinal canal stenosis (vertebral canal ratio = sagittal diameter of vertebral canal / sagittal diameter of vertebral body < 0.75).
5. Those suffering from severe heart, lung, brain, liver, kidney, or hematopoietic system diseases.
6. Conditions such as spinal tuberculosis, osteomyelitis, and osteoporosis.
7. Individuals who have undergone cervical spine surgery and those with cervical spine deformities.
8. Pregnant, planning to become pregnant, or breastfeeding women.
9. Participants unable to complete this clinical study due to mental illness, cognitive, or emotional disorders.
10. Those who have participated in other clinical studies in the past 3 months.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The Visual Analog Scale for Pain | 4 weeks
  The Visual Analog Scale for Pain is a tool used to assess the intensity of pain experienced by an individual. It consists of a straight line with "painless" marked at one end and "severe pain" at the other. The individual is asked to mark on the line the point that represents their current level of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain. The higher score indicates more severe pain.

SECONDARY OUTCOMES:
The Visual Analog Scale for Pain | 2 weeks
  The Visual Analog Scale for Pain is a tool used to assess the intensity of pain experienced by an individual. It consists of a straight line with "painless" marked at one end and "severe pain" at the other. The individual is asked to mark on the line the point that represents their current level of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain. The higher score indicates more severe pain.
The Visual Analog Scale for Pain | 8 weeks
  The Visual Analog Scale for Pain is a tool used to assess the intensity of pain experienced by an individual. It consists of a straight line with "painless" marked at one end and "severe pain" at the other. The individual is asked to mark on the line the point that represents their current level of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain. The higher score indicates more severe pain.
The Visual Analog Scale for Pain | 12 weeks
  The Visual Analog Scale for Pain is a tool used to assess the intensity of pain experienced by an individual. It consists of a straight line with "painless" marked at one end and "severe pain" at the other. The individual is asked to mark on the line the point that represents their current level of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain. The higher score indicates more severe pain.
The Visual Analog Scale for Pain | 16 weeks
  The Visual Analog Scale for Pain is a tool used to assess the intensity of pain experienced by an individual. It consists of a straight line with "painless" marked at one end and "severe pain" at the other. The individual is asked to mark on the line the point that represents their current level of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain. The higher score indicates more severe pain.
The Visual Analog Scale for Pain | 20 weeks
  The Visual Analog Scale for Pain is a tool used to assess the intensity of pain experienced by an individual. It consists of a straight line with "painless" marked at one end and "severe pain" at the other. The individual is asked to mark on the line the point that represents their current level of pain. Painless is represented by 0; 1-3 points represent mild pain; 4-6 points represent moderate pain, which is strong but tolerable; 7-10 points represent severe pain, gradually reaching intolerable level, which is severe pain. The higher score indicates more severe pain.
The Visual Analog Scale for Numbness | 2 weeks
  The Visual Analog Scale for Numbness is a tool used to assess the intensity of numbness experienced by an individual. It consists of a straight line with "unnumbness" marked at one end and "severe numbness" at the other. The individual is asked to mark on the line the point that represents their current level of numbness. Unnumbness is represented by 0; 1-3 points represent mild numbness; 4-6 points represent moderate numbness, which is strong but tolerable; 7-10 points represent severe numbness, gradually reaching intolerable level, which is severe numbness. The higher score indicates more severe numbness.
The Visual Analog Scale for Numbness | 4 weeks
  The Visual Analog Scale for Numbness is a tool used to assess the intensity of numbness experienced by an individual. It consists of a straight line with "unnumbness" marked at one end and "severe numbness" at the other. The individual is asked to mark on the line the point that represents their current level of numbness. Unnumbness is represented by 0; 1-3 points represent mild numbness; 4-6 points represent moderate numbness, which is strong but tolerable; 7-10 points represent severe numbness, gradually reaching intolerable level, which is severe numbness. The higher score indicates more severe numbness.
The Visual Analog Scale for Numbness | 8 weeks
  The Visual Analog Scale for Numbness is a tool used to assess the intensity of numbness experienced by an individual. It consists of a straight line with "unnumbness" marked at one end and "severe numbness" at the other. The individual is asked to mark on the line the point that represents their current level of numbness. Unnumbness is represented by 0; 1-3 points represent mild numbness; 4-6 points represent moderate numbness, which is strong but tolerable; 7-10 points represent severe numbness, gradually reaching intolerable level, which is severe numbness. The higher score indicates more severe numbness.
The Visual Analog Scale for Numbness | 12 weeks
  The Visual Analog Scale for Numbness is a tool used to assess the intensity of numbness experienced by an individual. It consists of a straight line with "unnumbness" marked at one end and "severe numbness" at the other. The individual is asked to mark on the line the point that represents their current level of numbness. Unnumbness is represented by 0; 1-3 points represent mild numbness; 4-6 points represent moderate numbness, which is strong but tolerable; 7-10 points represent severe numbness, gradually reaching intolerable level, which is severe numbness. The higher score indicates more severe numbness.
The Visual Analog Scale for Numbness | 16weeks
  The Visual Analog Scale for Numbness is a tool used to assess the intensity of numbness experienced by an individual. It consists of a straight line with "unnumbness" marked at one end and "severe numbness" at the other. The individual is asked to mark on the line the point that represents their current level of numbness. Unnumbness is represented by 0; 1-3 points represent mild numbness; 4-6 points represent moderate numbness, which is strong but tolerable; 7-10 points represent severe numbness, gradually reaching intolerable level, which is severe numbness. The higher score indicates more severe numbness.
The Visual Analog Scale for Numbness | 20 weeks
  The Visual Analog Scale for Numbness is a tool used to assess the intensity of numbness experienced by an individual. It consists of a straight line with "unnumbness" marked at one end and "severe numbness" at the other. The individual is asked to mark on the line the point that represents their current level of numbness. Unnumbness is represented by 0; 1-3 points represent mild numbness; 4-6 points represent moderate numbness, which is strong but tolerable; 7-10 points represent severe numbness, gradually reaching intolerable level, which is severe numbness. The higher score indicates more severe numbness.
The Neck Disability Index | 2 weeks
  The Neck Disability Index (NDI) is a widely used questionnaire designed to assess disability related to neck pain. It consists of ten items that evaluate different aspects of a person's daily activities and the impact of neck pain on their functionality. The NDI covers areas such as pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping, and recreation. Each item is scored on a scale from 0 to 5, with 0 indicating no disability and 5 indicating complete disability. The total score is then calculated by summing up the individual scores for each item, resulting in a possible range from 0 to 50. Higher scores on the NDI indicate greater disability and impairment due to neck pain.
The Neck Disability Index | 4 weeks
  The Neck Disability Index (NDI) is a widely used questionnaire designed to assess disability related to neck pain. It consists of ten items that evaluate different aspects of a person's daily activities and the impact of neck pain on their functionality. The NDI covers areas such as pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping, and recreation. Each item is scored on a scale from 0 to 5, with 0 indicating no disability and 5 indicating complete disability. The total score is then calculated by summing up the individual scores for each item, resulting in a possible range from 0 to 50. Higher scores on the NDI indicate greater disability and impairment due to neck pain.
The Neck Disability Index | 8 weeks
  The Neck Disability Index (NDI) is a widely used questionnaire designed to assess disability related to neck pain. It consists of ten items that evaluate different aspects of a person's daily activities and the impact of neck pain on their functionality. The NDI covers areas such as pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping, and recreation. Each item is scored on a scale from 0 to 5, with 0 indicating no disability and 5 indicating complete disability. The total score is then calculated by summing up the individual scores for each item, resulting in a possible range from 0 to 50. Higher scores on the NDI indicate greater disability and impairment due to neck pain.
The Neck Disability Index | 12 weeks
  The Neck Disability Index (NDI) is a widely used questionnaire designed to assess disability related to neck pain. It consists of ten items that evaluate different aspects of a person's daily activities and the impact of neck pain on their functionality. The NDI covers areas such as pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping, and recreation. Each item is scored on a scale from 0 to 5, with 0 indicating no disability and 5 indicating complete disability. The total score is then calculated by summing up the individual scores for each item, resulting in a possible range from 0 to 50. Higher scores on the NDI indicate greater disability and impairment due to neck pain.
The Neck Disability Index | 16 weeks
  The Neck Disability Index (NDI) is a widely used questionnaire designed to assess disability related to neck pain. It consists of ten items that evaluate different aspects of a person's daily activities and the impact of neck pain on their functionality. The NDI covers areas such as pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping, and recreation. Each item is scored on a scale from 0 to 5, with 0 indicating no disability and 5 indicating complete disability. The total score is then calculated by summing up the individual scores for each item, resulting in a possible range from 0 to 50. Higher scores on the NDI indicate greater disability and impairment due to neck pain.
The Neck Disability Index | 20 weeks
  The Neck Disability Index (NDI) is a widely used questionnaire designed to assess disability related to neck pain. It consists of ten items that evaluate different aspects of a person's daily activities and the impact of neck pain on their functionality. The NDI covers areas such as pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping, and recreation. Each item is scored on a scale from 0 to 5, with 0 indicating no disability and 5 indicating complete disability. The total score is then calculated by summing up the individual scores for each item, resulting in a possible range from 0 to 50. Higher scores on the NDI indicate greater disability and impairment due to neck pain.
The Short Form 12 | 2 weeks
  The Short Form 12 (SF-12) consists of 12 questions that cover various aspects of physical and mental health. It is designed to be a concise yet comprehensive measure of health status. The SF-12 questionnaire includes questions related to physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each question has multiple response options, and the responses are scored and aggregated to produce summary scores for physical health and mental health components. The SF-12 provides two main summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The total scores vary based on individual responses and can range from 0 to 100, with 100 representing the best possible health status and 0 representing the worst.
The Short Form 12 | 4 weeks
  The Short Form 12 (SF-12) consists of 12 questions that cover various aspects of physical and mental health. It is designed to be a concise yet comprehensive measure of health status. The SF-12 questionnaire includes questions related to physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each question has multiple response options, and the responses are scored and aggregated to produce summary scores for physical health and mental health components. The SF-12 provides two main summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The total scores vary based on individual responses and can range from 0 to 100, with 100 representing the best possible health status and 0 representing the worst.
The Short Form 12 | 8 weeks
  The Short Form 12 (SF-12) consists of 12 questions that cover various aspects of physical and mental health. It is designed to be a concise yet comprehensive measure of health status. The SF-12 questionnaire includes questions related to physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each question has multiple response options, and the responses are scored and aggregated to produce summary scores for physical health and mental health components. The SF-12 provides two main summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The total scores vary based on individual responses and can range from 0 to 100, with 100 representing the best possible health status and 0 representing the worst.
The Short Form 12 | 12 weeks
  The Short Form 12 (SF-12) consists of 12 questions that cover various aspects of physical and mental health. It is designed to be a concise yet comprehensive measure of health status. The SF-12 questionnaire includes questions related to physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each question has multiple response options, and the responses are scored and aggregated to produce summary scores for physical health and mental health components. The SF-12 provides two main summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The total scores vary based on individual responses and can range from 0 to 100, with 100 representing the best possible health status and 0 representing the worst.
The Short Form 12 | 16 weeks
  The Short Form 12 (SF-12) consists of 12 questions that cover various aspects of physical and mental health. It is designed to be a concise yet comprehensive measure of health status. The SF-12 questionnaire includes questions related to physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each question has multiple response options, and the responses are scored and aggregated to produce summary scores for physical health and mental health components. The SF-12 provides two main summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The total scores vary based on individual responses and can range from 0 to 100, with 100 representing the best possible health status and 0 representing the worst.
The Short Form 12 | 20 weeks
  The Short Form 12 (SF-12) consists of 12 questions that cover various aspects of physical and mental health. It is designed to be a concise yet comprehensive measure of health status. The SF-12 questionnaire includes questions related to physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each question has multiple response options, and the responses are scored and aggregated to produce summary scores for physical health and mental health components. The SF-12 provides two main summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The total scores vary based on individual responses and can range from 0 to 100, with 100 representing the best possible health status and 0 representing the worst.
The total cost | 4 weeks
  The total cost includes registration fees, treatment fees, examination fees, loss of income, transportation expenses, and so on. Record the total costs for each group of patients over a 4-week treatment period.
The recurrence rate | 20 weeks
  The recurrence rate is defined as the percentage of individuals experiencing a reappearance of symptoms and signs similar to those before treatment during the follow-up period, among the total number of revisit cases.
Expectation of Treatment and Credibility Scale | 1 day
  The Expectation of Treatment and Credibility Scale (ETCS) is a questionnaire commonly used in clinical practice to assess patients' expectations of treatment outcomes and their perceived credibility of the treatment. Responses on the ETCS are usually rated on a Likert 9-point scale (from 0 to 9), with options ranging from "strongly disagree" to "strongly agree" or "not at all credible" to "extremely credible." Scores are then calculated to provide quantitative measures of patients' expectations and perceived credibility of the treatment. Overall, higher ETCS scores generally indicate higher patient expectations for treatment options and greater trust in treatment. This may help improve the effectiveness of treatment and patient satisfaction. Evaluation was performed after the first treatment and at 4 weeks of treatment.
Expectation of Treatment and Credibility Scale | 4 weeks
  The Expectation of Treatment and Credibility Scale (ETCS) is a questionnaire commonly used in clinical practice to assess patients' expectations of treatment outcomes and their perceived credibility of the treatment. Responses on the ETCS are usually rated on a Likert 9-point scale (from 0 to 9), with options ranging from "strongly disagree" to "strongly agree" or "not at all credible" to "extremely credible." Scores are then calculated to provide quantitative measures of patients' expectations and perceived credibility of the treatment. Overall, higher ETCS scores generally indicate higher patient expectations for treatment options and greater trust in treatment. This may help improve the effectiveness of treatment and patient satisfaction. Evaluation was performed after the first treatment and at 4 weeks of treatment.
Adverse reactions | Up to 20 weeks
  Recording whether patients experience adverse reactions such as progressive worsening of neck pain, upper limb pain, and restricted neck movement, dizziness, chest tightness, palpitations, etc., during the treatment and follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Wangjing Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The researchers do not currently plan to share IPD. Our team is also conducting some other studies on the rotation-traction manipulation. We will consider disseminating our data more openly after the results of these studies are published. However, if other researchers are interested in our research, they can contact the author team to obtain relevant information. Let's work together to contribute to the international dissemination of traditional Chinese medical manipulations.

REFERENCES:
- [Background] Bono CM, Ghiselli G, Gilbert TJ, Kreiner DS, Reitman C, Summers JT, Baisden JL, Easa J, Fernand R, Lamer T, Matz PG, Mazanec DJ, Resnick DK, Shaffer WO, Sharma AK, Timmons RB, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of cervical radiculopathy from degenerative disorders. Spine J. 2011 Jan;11(1):64-72. doi: 10.1016/j.spinee.2010.10.023. PMID 21168100